CLINICAL TRIAL: NCT02368509
Title: Sensory Approach of Food Modifications Led by Chemotherapy
Acronym: ARC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014.871; 2014-A00742-45 (Other: ANSM)
Record Dates: First submitted 2014-12-05; First posted 2015-02-23 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: sensory test; olfaction; gustation; taste; cancer
MeSH Terms: conditions — Neoplasms; Anosmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bronchial cancer (Experimental): Patients with bronchial cancer will perform sensory tests before and after a 6-week period of chemotherapy.
  Interventions: Other: Perform sensory tests
- Control group (Placebo Comparator): Healthy individuals will perform sensory tests before and after a 6-week period without chemotherapy.
  Interventions: Other: Perform sensory tests

INTERVENTIONS:
Other: Perform sensory tests

SUMMARY:
The aim of the present study was to evaluate the impact of chemotherapy on sensorial perception in lung cancer patients in comparison to a control group (individuals without lung cancer and chemotherapy treatment). We will use a longitudinal approach whereby 44 patients and 44 controls will be tested for olfactory and gustatory abilities before and after treatment (for patients) and for two sessions separated by the same duration for controls. Primary measure outcome will be to examine the impact of treatment on the perception of hedonic valence of odors. Secondary measure outcome will include odor and taste perceptual changes and questionnaires on eating habits and behaviors, in order to examine the impact of treatment on odor, taste and food perception.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age ≥ 18 years old
* People capable of giving their consent and of understanding the study
* 18 ≤ BMI < 30 kg/m²

Control group:

* controlled blood pressure
* absence of pathology which can interfere with the criteria of the study (ENT, neurological, digestive,…)
* absence of treatment which can interfere with the criteria of the study
* absence of digestive disorders
* women with contraception

Patients:

* Patients affected by a bronchial cancer (post-operative or metastatic) with small cells or not, that must be handled by a chemotherapy with salts of platinum (at least 3 cycles)
* patients without previous chemotherapy
* Absence of ENT or neurological pathologies

Exclusion Criteria:

- Subjects having lost more than 10 % of their weight in the previous 2 months

Patients:

* Symptomatic intellectual and/or meningeal metastases
* Mycosis of oral or superior digestive tract
* Cancer of ENT or esophageal or gastric ways
* Patients with digestive disorders (≥ rank 1)
* Patients presenting a pathology which can interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Change in Pleasantness judgments in the European Test of Olfactory Capabilities (ETOC) | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  Fed state This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (very unpleasant) to 9 (very pleasant).

SECONDARY OUTCOMES:
Change in Intensity judgment (IJ-ETOC) of odors in the ETOC test | Before (day 1) and after the 6-week period (day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (no odor) to 9 (very intense odor).
Change in Intensity judgment (IJ-8odor) of odors in the 8-odor test | Before (day 1) and after the 6-week period (day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (no odor) to 9 (very intense odor).
Change in Intensity judgment (IJ-Taste) of tastes in the Taste Strips test | Before (day 1) and after the 6-week period (day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (no taste) to 9 (very intense taste).
Change in Familiarity judgment (FJ-ETOC) of odors in the ETOC test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (unknown odor) to 9 (very known odor).
Change in Familiarity judgment (FJ-8odor) of odors in the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (unknown odor) to 9 (very known odor).
Change in Familiarity judgment (FJ-Taste) of tastes in the Taste Strips test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (unknown taste) to 9 (very known taste).
Change in Edibility judgment (EJ-ETOC) of odors in the ETOC test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (not edible) to 9 (very edible).
Change in Edibility judgment (EJ-8odor) of odors in the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (not edible) to 9 (very edible).
Change in Pungency judgments (PUJ) of odors for the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (not at all pungent) to 9 (very pungent).
Change in Warmness judgments (WAJ) of odors for the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (not at all warm) to 9 (very warm).
Change in Coolness judgments (COJ) of odors for the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (not at all cool) to 9 (very cool).
Change in Irritation judgments (IRJ) of odors for the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (not at all irritant) to 9 (very irritant).
Change in Olfactory detection (OD-ETOC) with the ETOC test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A score from 0 (no odor detected) to 16 (all odors detected) is collected.
Change in Olfactory identification (OI-ETOC) in the ETOC test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure:A score from 0 (no odor identified) to 16 (all odors identified) is collected.
Change in Olfactory identification (OI) in the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A score from 0 (no odor identified) to 8 (all odors identified) is collected.
Change in Gustatory detection (GD) in the Taste Strips test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: a score from 0 (no taste detected) to 4 (all tastes detected) is collected.
Change in Gustatory identification (GI) in the Taste Strips test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: a score from 0 (no taste identified) to 4 (all tastes identified) is collected.
Change in Pleasantness judgment (PJ-8odor) of odors in the 8-odor test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (very unpleasant odor) to 9 (very pleasant odor).
Change in Pleasantness judgment (PJ-Taste) of tastes in the Taste Strips test | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  This score will be evaluated before and after a 6-week period (i) of chemotherapy for patients with bronchial cancer and (ii) without chemotherapy for control subjects.
  Unit of measure: A visual scale is used to collect a score from 1 (very unpleasant taste) to 9 (very pleasant taste).
practices and food habits | Before (Day 1) and after treatment (Day 42) - (On average 3 weeks and 9 weeks after patient's inclusion)
  Practices and food habits will be evaluated before and after the 6-week period. Food odors which appeared less or more agreeable the weeks before the survey will also be evaluated before and after the 6-week period.
  Unit of measure: these measures are qualitative; the results will be expressed in percentage of given responses.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre de Recherche en Nutrition Humaine, Pierre-Bénite
  - Centre Hospitalier Lyon Sud - Service de Pneumologie, Pierre-Bénite
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Result] Drareni K, Dougkas A, Giboreau A, Laville M, Souquet PJ, Nazare JA, Fournel P, Bensafi M. Loss of smell in lung cancer patients undergoing chemotherapy: Prevalence and relationship with food habit changes. Lung Cancer. 2023 Mar;177:29-36. doi: 10.1016/j.lungcan.2023.01.007. Epub 2023 Jan 12. PMID 36701841
- See also: Related Info — https://www.crnh-rhone-alpes.fr/
- See also: Related Info — http://recherche.institutpaulbocuse.com/
- See also: Related Info — http://crnlgerland.univ-lyon1.fr